CLINICAL TRIAL: NCT00313066
Title: Comparison the Level of CTGF Protein and Related Cytokine in Pleural Effusion Among Tuberculous Pleurisy and Malignant Pleural Effusion Patients
Brief Title: Comparison the Level of CTGF Protein and Related Cytokine in Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Ton General Hospital (Unknown)
Other Study IDs: 940513/C05092
Record Dates: First submitted 2006-04-09; First posted 2006-04-11 (Estimated); Last update posted 2006-04-11 (Estimated); Status verified 2006-04

CONDITIONS: Tuberculosis; Tuberculous Pleurisy; Malignant Pleural Effusion; Empyema
Keywords: CTGF; fibrogenic cytokine; FGF; pleural fibrosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pleural; Pleural Effusion, Malignant; Empyema

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Connective tissue growth factor (CTGF) is known to be a fibrogenic cytokine, it could be expressed in various fibrosis diseases. But, recent research showed that CTGF also be considered to be a tumor suppressive gene. The expression of CTGF protein is higher in normal Type I and II alveolar epithelial cells than metastatic tumor cells. CTGF appears to be a suppressor of lung tumor invasion and in metastasis and the decreased CTGF expression in tumor tissues was associated with advanced tumor stage, lymph node metastasis, early postoperative relapse and shorter patient survival.

CTGF can be expressed in many human organs such as heart, brain, placenta, liver, muscle, kidney, peritoneal mesothelial cells and lung but did not known in the pleura. The CTGF protein is present in the peritoneal cavity and is increased during peritonitis. Considering pleural cavity comes from the same origin of mesenchyma with peritoneum, pericardium and fallopian tube, we aim to evaluate whether the CTGF expression increase in the pleurisy patients including the parapneumonic effusion and the TB pleurisy.

The diagnosis of TB pleurisy depends on the effusion TB culture and pleural biopsy. Unfortunately the sensitivity of TB culture was only 20-30%. So most patients must receive invasive pleural biopsy. Adenosine deaminase(ADA) was developed as a screening test but should not be considered an alternative test to culture and biopsy. The sensitivity of ADA might vary from 32%-100% and the cutoff value also vary from 26 to 70 IU/L. We should develop a method to alternate the culture and biopsy . Therefore, our technologist Jao-Jia chu will develop the CTGF ELISA kit for this specific aim. If CGTF might increase expression in pleuritis but decrease in pleural metastasis, it might be a potential method help to differentiate lymphocytic pleural effusion between TB pleurisy and malignancy.

DETAILED DESCRIPTION:
Connective tissue growth factor (CTGF, also known as CCN2) is a member of the CCN family. Cysteine-rich 61(Cyr61) is known as CCN1, and nephroblastoma over-expressed (Nov, known as CCN3) as well as Wisp-1/elm1( CCN4),Wisp-2/rCop1(CCN5), and Wisp-3 (CCN6)1. The CTGF is a secretory growth factor that bind with integrins on the cell surface and was first identified as a mitogen isolated from the medium of human umbilical vein endothelial cells2. CTGF can be expressed in many human organs such as heart, brain, placenta, liver, muscle, kidney, and lung and may have many biologic functions3. CTGF stimulate the proliferation of fibroblast and vascular endothelial cells. The level of CTGF protein is increased in patients with various fibrotic human disease including renal failure, hepatic fibrosis in biliary atresia, systemic scleroderma and vascular atherosclerosis4.

Recent research revealed the expression of CTGF protein was high in the normal lung epithelium and moderate to high in stage I lung adenocarcinoma cells5. But the expression of CTGF was reduced in low grade metastatic respiratory epithelial tumor cells. The CTGF expression was associated with the suppression of human lung cancer cell metastasis in a mouse model and the reduced CTGF expression was also associated with clinical metastasis and patient survival5. The expression of CTGF protein was statistically significantly higher in normal lung type I and II epithelial cells than in the majority of metastatic adenocarcinoma specimens revealed that the level of CTGF protein decreases during clinical disease when cells acquire the ability to grow at metastatic site6. CTGF appears to be a suppressor of lung tumor invasion and metastasis and the decreased CTGF expression in tumor tissues was associated with advanced tumor stage, lymph node metastasis, early postoperative relapse, and shorter patient survival. Connective tissue growth factor acts as an independent prognostic marker in colorectal cancer and giomas and inhibits metastasis7,8

ELIGIBILITY:
Inclusion Criteria:

- patients with pleural effusion

Exclusion Criteria:

* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-11; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Shen Gwan Han, MD, Principal Investigator — Division of Chest Medicine, Department of Internal Medicine, Taichung Veterans General Hospital
Locations (1):
- Division of Chest Medicine, Department of Internal Medicine, Taichung Veterans General Hospital, Taichung, Taiwan, China